CLINICAL TRIAL: NCT05864391
Title: A Phase I Randomized Single-blind Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD7503 Following Multiple Ascending Dose Administration to Patients With Suspected Non-cirrhotic Non-alcoholic Steatohepatitis (NASH)
Brief Title: A Study to Investigate Safety, Tolerability, and Pharmacokinetics of AZD7503 in Participants With Suspected NASH.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: AstraZeneca have decided to not move forward with the development of the compound.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: D9230C00002
Record Dates: First submitted 2023-04-20; First posted 2023-05-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Steatohepatitis
Keywords: Cirrhosis
MeSH Terms: conditions — Fatty Liver; Fibrosis

STUDY DESIGN:
Intervention Model Description: Each participant is expected to be in the study for approximately 24 weeks, including a screening period of up to 4 weeks, a 12-week study intervention period, and a follow-up visit at week 18 (10 weeks following the final dose). Participants will be randomly assigned in a 3:1 ratio to receive AZD7503 or placebo. Study intervention will be administered via subcutaneous injection.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a single-blind, randomised, placebo-controlled, MAD study with up to 3 study intervention cohorts that are participant- and investigator-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Other): Dose A cohort: 20 participants; n=15 on AZD7503 dose A, n=5 on Placebo
  Interventions: Drug: AZD7503
- Cohort 2 (Other): Dose B cohort: 20 participants; n=15 on AZD7503 dose B, n=5 on Placebo.
  Interventions: Drug: AZD7503
- Cohort 3 (Other): Dose C cohort: 20 participants n=15 on AZD7503 dose C, n=5 on Placebo.
  Interventions: Drug: AZD7503

INTERVENTIONS:
Drug: AZD7503 — Each participant is expected to be in the study for approximately 24 weeks, including a screening period of up to 28 days, a 12-week study intervention period, and a follow-up visit at week 18 (10 weeks following the final dose). Participants will be randomly assigned in a 3:1 ratio to receive AZD7503 or placebo. Study intervention will be administered via subcutaneous injection.

SUMMARY:
The purpose of this study is to measure the safety, tolerability, and PK (measurement of drug activity in the body over time) of AZD7503 injected subcutaneously, and compared to placebo, in participants with suspected NASH, a type of liver disease.

DETAILED DESCRIPTION:
This is a Phase I, randomised, single-blind (in which the study centre staff including the Principal Investigator, remain blinded during the clinical conduct of a given cohort) placebo controlled, multiple ascending dose (MAD) study in male and female participants conducted at multiple centres.

Each participant is expected to be in the study for approximately 24 weeks, including a screening period of up to 4 weeks, a 12-week study intervention period, and a follow-up visit at week 18 (10 weeks following the final dose). Participants will be randomly assigned in a 3:1 ratio to receive AZD7503 or placebo. Study intervention will be administered via subcutaneous injection.

ELIGIBILITY:
Key Inclusion Criteria

1. Biopsy-confirmed NASH diagnosis with CRN score of fibrosis stage of F1 to F3 within the previous 12 months prior to screening or history of fatty liver disease by imaging plus clinical suspicion of NASH based on history of type 2 DM for at least 5 years or overweight/obesity with BMI 25 to 40 kg/m^2 with 2 additional metabolic syndrome components.
2. Males and females of non-child bearing potential.
3. Willing to provide written informed consent and comply with study requirements.

Key Exclusion Criteria

1. Evidence of any clinical important condition which in the investigator opinion makes it undesirable for the participant to participate in the study
2. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention
3. History of liver transplant or presence or history of hepatic disease other than NASH or histological or imaging evidence of cirrhosis.
4. Human immunodeficiency virus (HIV) infection, seropositive for Hepatitis B (HBV)virus, seropositive for Hepatitis C virus (HCV)
5. History of excessive alcohol consumption
6. Uncontrolled high blood pressure
7. Any clinically important abnormalities in ECG
8. Suspected history of illicit drug abuse
9. Clinically important abnormalities in urine and blood laboratory results
10. Changes in concomitant medication within 1 month of screening
11. Received another investigational drug within 90 days of administration of study intervention in this study
12. Has received any chemical entity or investigational drug targeting HSD17B13 (eg, ARO-HSD or ALN-HSD).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) | Up to and including week 19 (from pre-screening to follow-up visit)
  AEs will be collected at all sites visits per SOA.
Number of subjects with serious adverse events (SAEs) | Up to and including week 18 (from pre-screening to final visit).
  SAEs will be reported and collected as they occur.

SECONDARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | Day 1 to Day 127
  PK parameters to be collected per the SOA.
Area under the concentration-time curve from time 0 to infinity (AUCinf) for plasma PK | Day 1 to 127
  PK parameters to be collected per the SOA.
Area under the concentration-time curve over the dosing interval (AUCtau) for plasma PK | Time frame: Day 1 to 127
  PK parameters to be collected per the SOA.
Fraction of the dose excreted unchanged into the urine from time t1 to t2 (fe(t1-t2)) for urine PK | Day 1 and Day 57: Pre-dose and between 0-6 hours, 6-12 hours, 12-24 hours, 24-36 hours and 36-48 hours post-dose
  PK parameters to be collected per the SOA.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - Research Site, Chandler, Arizona
  - Research Site, Montclair, California
  - Research Site, Hialeah, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Morehead City, North Carolina
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
- Research Site, San Juan, Puerto Rico

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9230C00002&attachmentIdentifier=31b28cb3-75eb-4f27-8cc0-ac91f5f3c646&fileName=D9230C00002_redacted_CSR_synopsis.pdf&versionIdentifier=